CLINICAL TRIAL: NCT06108401
Title: Effect Of a Goat Milk-Based Infant Formula On Gastrointestinal And Other Symptoms And Health-Related Quality Of Life.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GMF-2023
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Infant Nutrition Disorders; Gastrointestinal Diseases
Keywords: goat milk; infant formula; nutrition
MeSH Terms: conditions — Infant Nutrition Disorders; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goat milk formula-fed group (Experimental): 79 participants
  Interventions: Dietary Supplement: Goat milk-based infant formula
- Cow milk formula-fed group (Placebo Comparator): 79 participants
  Interventions: Dietary Supplement: Cow milk-based infant formula

INTERVENTIONS:
Dietary Supplement: Goat milk-based infant formula — Goat milk-based infant formula exclusively for 4 weeks at a volume depending on the infant.
  Arms: Goat milk formula-fed group
Dietary Supplement: Cow milk-based infant formula — Regular cow milk-based infant formula that is similar in color, smell, and taste to the formula received by the experimental group.
  Arms: Cow milk formula-fed group

SUMMARY:
In this trial, the investigators aim to assess impact of goat milk-based infant formula on the severity and frequency of gastrointestinal symptoms, as well as other associated symptoms, and the health-related quality of life in infants exhibiting symptoms possibly related to cow's milk, compared to a cow milk-based formula.

DETAILED DESCRIPTION:
Gastrointestinal symptoms are frequent in the first 6 months of life in otherwise healthy infants fed cow milk-based infant formulas (CMF). In management special infant formulas may be considered, although none is routinely recommended. Goat milk-based infant formulas (GMF) have shown promising effects on digestion and increased gastric emptying in several in vitro studies.

In this trial, a total of 158 participants at age 14 to 90 days, who exhibit gastrointestinal and/or other symptoms associated with CMF consumption, as assessed with the Cow's Milk-related Symptom Score (CoMiSS) between 6 and 10 will be randomly allocated to GMF or CMF for four weeks. The primary outcome will be the proportion of infants showing a reduction of at least 4 points in CoMiSS following the four-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants with a gestational age between 37 and 42 weeks.
* Infants who have received cow's milk infant formula for at least 7 consecutive days.
* Exclusive formula feeding.
* Cow's Milk-related Symptoms Score (CoMiSS) value at baseline between ≥6 and <10.

Exclusion Criteria:

* exclusive or partial breastfeeding (or feeding human milk)
* introduced to solid food/supplementary feeding
* any congenital or chronic condition
* previous or present gastrointestinal illness or malformation that could interfere with study parameters
* diagnosed cow's milk allergy
* receiving medication with regard to functional gastrointestinal disorders (i.e., reflux medication)
* sibling already participating in this study, and/or participating in another clinical trial.

Ages: 14 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of Cow's Milk-related Symptoms Score (CoMiSS) values after 4 weeks | 0 - 4 weeks
  Proportion of infants with a reduction of 4 points or more in the CoMiSS value

SECONDARY OUTCOMES:
Reduction of Cow's Milk-related Symptoms Score (CoMiSS) values after 2 weeks | 0 - 2 weeks
  Proportion of infants with a reduction of 4 points or more in the CoMiSS value
Difference in Cow's Milk-related Symptoms Score (CoMiSS) values after 2 weeks | 0 - 2 weeks
  Difference in the CoMiSS between infants fed with goat milk-based infant formula versus cow milk-based infant formula
Difference in Cow's Milk-related Symptoms Score (CoMiSS) values after 4 weeks | 0 - 4 weeks
  Difference in the CoMiSS between infants fed with goat milk-based infant formula versus cow milk-based infant formula
The Pediatric Quality of Life Inventory (PedsQL) Infant Scales improvement after 2 weeks | 0 - 2 weeks
  Proportion of infants with a PedsQL Infant Scale score of 80 or higher
The Pediatric Quality of Life Inventory (PedsQL) Infant Scales improvement after 4 weeks | 0 - 4 weeks
  Proportion of infants with a PedsQL Infant Scale score of 80 or higher
Improvement in gastrointestinal symptoms measured by the Infant Gastrointestinal Symptom Questionnaire (IGSQ) after 2 weeks | 0 - 2 weeks
  Change in the severity and frequency of gastrointestinal symptoms as measured by the IGSQ
Improvement in gastrointestinal symptoms measured by the Infant Gastrointestinal Symptom Questionnaire (IGSQ) after 4 weeks | 0 - 4 weeks
  Change in the severity and frequency of gastrointestinal symptoms as measured by the IGSQ
Anthropometric parameters after 2 weeks | 0 - 2 weeks
  Assessment of growth parameters, including weight
Anthropometric parameters after 4 weeks | 0 - 4 weeks
  Assessment of growth parameters, including weight
Adverse events | 0 - 4 weeks
  Adverse events throughout the study period
Anthropometric parameters after 2 weeks | 0 - 2 weeks
  Assessment of growth parameters, including length
Anthropometric parameters after 4 weeks | 0 - 4 weeks
  Assessment of growth parameters, including length

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Jankiewicz, MD, Principal Investigator — Department of Paediatrics, The Medical University of Warsaw, Poland
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw, Poland